CLINICAL TRIAL: NCT01762826
Title: Adverse Obstetric Outcomes in Gestational Diabetes Mellitus and Inositol Stereoisomears
Brief Title: Myo-inositol, D-chiro-inositol, and D-chiro/Myo-inositol in Gestational Diabetes
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: G. d'Annunzio University (Other)
Collaborators: University of Chieti (Other)
Responsible Party: Principal Investigator, Claudio Celentano, MD, G. d'Annunzio University
Other Study IDs: INOS002
Record Dates: First submitted 2012-11-25; First posted 2013-01-08 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2012-09

CONDITIONS: GDM
Keywords: Inositol; GDM
MeSH Terms: interventions — Inositol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Placebo control: Diet pills of 400 mcg of acid folic daily
  Interventions: Dietary Supplement: Placebo
- D-chiro-inositol / Myo-inositol: Diet sachets 2000 mg myo-inositol and 250 mg d-chiro-inositol and 400 mcg folic acid daily
  Interventions: Dietary Supplement: D-Chiro / Myo-inositol
- D-chiro-inositol: Diet pills with 500 mg d-chiro-inositol and 400 mcg folic acid daily
  Interventions: Dietary Supplement: D-chiro-inositol
- Myo-inositol: Diet sachets with 2000 mg myo-inositol and 200 mcg folic acid twice daily
  Interventions: Dietary Supplement: Myo-inositol

INTERVENTIONS:
Dietary Supplement: Myo-inositol — Dietary control plus Myo-inositol
  Other Names: Supplementation of myo-inositol plus dietary control
  Groups: Myo-inositol
Dietary Supplement: D-chiro-inositol — Dietary control plus D-Chiro-Inositol supplementation
  Groups: D-chiro-inositol
Dietary Supplement: D-Chiro / Myo-inositol — Dietary control Supplementation with myo and d-chiro inositol
  Groups: D-chiro-inositol / Myo-inositol
Dietary Supplement: Placebo — Dietary control plus folic acid 400 mcg daily
  Groups: Placebo control

SUMMARY:
Comparison of different inositol stereoisomears in preventing adverse obstetric outcomes in non-obese pregnant women at high risk for gestational diabetes mellitus.

DETAILED DESCRIPTION:
The investigators compared outcomes from metabolic and obstetric point of view in GDM pregnant non-obese patient with different stereoisomears of inositol supply. Dietary control and placebo or inositol steroisomears were administered starting at the enrolling time (first fasting oral glucose above 92 mg%; usually before 20 weeks gestations') till the delivery and/or pregnancy end/termination. Oral glucose tolerance test results at 24-28 weeks' gestation was evaluated (as glucose values and oGTT screening). Fetal growth, delivery data, obstetric outcomes and necessity of insulin therapy were taken into account.

ELIGIBILITY:
Inclusion Criteria:

* pregnancy below 20 weeks gestation BMI below 30 Fasting glucose between 92 and 126 mg% Singleton pregnancy Naturally conceived

Exclusion Criteria:

* obese patient Fasti g glucose above 126 or below 92

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Non obese pregnant women during first trimester of pregnancy with scared fasting glucose (above 92 mg%)
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2012-09; Primary Completion 2013-04 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
OGTT result | 24-28 weeks' gestation
  OGTT is the mainstay of obstetric outcomes in GDM

SECONDARY OUTCOMES:
Fetal measurements at third trimester | 28 weeks
  Centiles of fetal measurements and amniotic fluid volume
Delivery data | 25-42 weeks gestations'
  Gestational age at delivery Route of delivery Fetal gender Fetal weight (grams and centiles) Neonatal hypoglycemia
Adverse obstetric outcome | from first elevated oral fasting glucose (above 92 mg%) till the end/termination of pregnancy (latter 42 weeks gestation)
  Abortion Preterm delivery Polyhydramnios IUGR Macrosomia Fetal distress Preterm delivery pPROM Neonatal morbility (NICU stay, low glucose levels, etc.) Neonatal mortality Cerebral palsy Route of delivery Dystocia Etc.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Celentano, MD, Study Director — ObGyn Dept University of Chieti; Barbara Matarrelli, MD, Principal Investigator — ObGyn Dept Univ of Chieti; Ester Vitacolonna, MD, Study Chair — Diabetology Dept Univ of Chieti